CLINICAL TRIAL: NCT06765746
Title: Repolarization and Activation Mapping in Ventricular Tachycardia Ablation: the REDEMPTION Study
Acronym: REDEMPTION
Status: Not yet recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Carlo de Asmundis, Head of the department: Heart Rhythm Management Centre, Postgraduate Course in Cardiac Electrophysiology and Pacing, Vrije Universiteit Brussel, Universitair Ziekenhuis, Universitair Ziekenhuis Brussel
Other Study IDs: REDEMPTION
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Ventricular Tachycardia Ablation
Keywords: ventricular tachycardia; EAM; Electroanatomical map; Substrate ablation; Catheter ablation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing ventricular tachycardia ablation: The intervention is standard of care. Ventricular tachycardia (VT) ablation will be performed following standard of care in all 40 patients in the arm. No experimental tool or comparator will be used.
  The study aims at evaluating a novel sinus rhythm mapping strategy. Furthermore, gathering clinical data on VT ablation with TactiFlex is also aimed. We aim at prospectively enrolling 40 patients in 1 year and to complete 1 year follow-up.
  Interventions: Procedure: Ventricular tachycardia ablation

INTERVENTIONS:
Procedure: Ventricular tachycardia ablation — All ventricular tachycardia (VT) ablation procedures will be performed under general anesthesia. An epicardial approach will be performed, if clinically needed, when a detailed endocardial mapping during VT fails to reveal the complete VT critical isthmus. In case of epicardial mapping, the pericardium will be accessed percutaneously using the method described by Sosa et al.
  VT activation mapping will be performed and the critical isthmus will be defined as the diastolic pathway.
  Ablation will be performed at 50 W (temperature limit of 43 °C) using an irrigated ablation catheter (TactiFlex, Abbott, MN). Ablation will be aimed at VT isthmus transection. Substrate modification will be added if the patient is still inducible or in the absence of any inducible/tolerated VT. Substrate ablation will be performed based on sinus rhythm mapping, aiming at non-inducibility of any VT. At the end of procedure, programmed ventricular stimulation will be repeated.

SUMMARY:
The aim of this study is to prospectively evaluate a novel sinus rhythm mapping strategy for ventricular tachycardia (VT) ablation based on combined ventricular repolarization and activation (depolarization) mapping (REpolarization DEpolarization Mapping, REDEEM mapping). Furthermore, gathering clinical data on VT ablation with TactiFlex is also aimed.

DETAILED DESCRIPTION:
INTRODUCTION Among therapeutic strategies for ventricular tachycardia (VT), catheter ablation is indicated in reducing ICD shocks, improving quality of life and survival in selected cases, such as arrhythmic storm. However, clinical outcomes of VT ablation are hampered by not hemodynamically tolerated VTs in up to 30% of cases or not inducible/sustained VTs1. In this setting, substrate mapping during sinus rhythm is of utmost importance to guide ablation in the absence of a mapped reentry circuit.

Since slow conduction and unidirectional block are necessary for any reentrant arrhythmia, most of sinus rhythm approaches are based on slow and late wavefront conduction such as: late potentials (LPs), local abnormal ventricular activities (LAVAs) and isochronal late activation maps (ILAM). However, for reentry to occur, the returning wavefront needs to occur with a timing compatible with the recovery of the repolarization in the upfront tissue (wave tail). Based upon these premises, recently, novel strategies based on repolarization (or wave tail) have also been assessed.

Human VT reentry circuit is arguably the result of an interplay between both a delayed conduction and repolarization heterogeneities. Thus, a substrate mapping method evaluating slow conduction together with repolarization abnormalities may capture the complexity of the reentrant VT phenomenon.

METHODOLOGY INCLUSION AND EXCLUSION CRITERIA All consecutive patients undergoing VT ablation at Universitair Ziekenhuis Brussel (UZB), Brussels, Belgium will be prospectively enrolled if inclusion criteria will be fulfilled. Inclusion criteria will be: 1) VT ablation procedure; 2) High density endocardial or epicardial substrate EAM performed with the multipolar mapping catheter Advisor™ HD-Grid Mapping Catheter, (Abbott Labs, Abbott Park, IL, USA) in association with the EnsiteXTM Cardiac Mapping System, (Abbott Labs, Abbott Park, IL, USA); 3) Use of TactiFlexTM ablation catheter (Abbott Labs, Abbott Park, IL, USA).

Exclusion criteria will be: 1) use of a different EAM mapping system. Clinical VT will be defined as a VT that occurs spontaneously based on analysis of 12-lead ECG QRS morphology, following current guidelines. Sustained VT will be defined as lasting more than 30 s. All patients will sign an informed consent. All data will be collected and updated in a centralized online database. The study will comply with the Declaration of Helsinki; the ethic committee will approve the study.

VENTRICULAR TACHYCARDIA MAPPING AND ABLATION All VT ablation procedures will be performed under general anesthesia. Antiarrhythmic drugs will be discontinued at least 5 half-lives before the procedure. An epicardial approach will be performed, if clinically needed, when a detailed endocardial mapping during VT fails to reveal the complete VT critical isthmus. In case of epicardial mapping, the pericardium will be accessed percutaneously using the method described by Sosa et al. Epicardial mapping will be performed after pericardial access, then systemic anticoagulation will be achieved by intravenous heparin with an activation clotting time of 250 to 350 s.

VT activation mapping will be performed and the critical isthmus will be defined as the diastolic pathway, following current guidelines. Diastolic potentials unrelated to the critical isthmus (i.e.: dead-end pathways and adjacent bystanders) will be ruled out after careful review and interpretation of the activation map or with entrainment mapping, if indicated. Mapping of a macroreentrant VT will be considered complete, as previously described, when: (1) ≥90% of the VT cycle lenght is mapped; (2) a diastolic channel of conduction isthmus is identified. Macroreentrant VT circuit components will be defined as follows: 1) Entrance site: the entrance will be defined as the site at which the orthodromic wavefront enters to the diastolic pathway; 2) Common diastolic pathway (mid-isthmus) and 3) Exit site: the exit site will be defined as the site at which the orthodromic wave front exits the common diastolic pathway.

All VT and substrate maps will be analyzed offline by two independent physicians. Discrepancies will be adjudicated by a third independent physician. Ablation will be performed at 50 W (temperature limit of 43 °C) using an irrigated ablation catheter (TactiFlex, Abbott, MN). Ablation will be aimed at VT isthmus transection. Substrate modification will be added if the patient is still inducible or in the absence of any inducible/tolerated VT. Substrate ablation will be performed based on sinus rhythm mapping, aiming at non-inducibility of any VT. At the end of procedure, programmed ventricular stimulation will be repeated up to four extrastimuli to confirm non-inducibility of any VT.

HIGH DENSITY SINUS RHYTHM ELECTROANATOMIC MAPPING AND ANALYSIS Electroanatomical maps will be created in sinus rhythm with a multielectrode high-density catheter Advisor™ HD-Grid Mapping Catheter, (Abbott Labs, Abbott Park, IL, USA). All maps will be performed during sinus rhythm with (1) intrinsic QRS activation when possible, or (2) right ventricular pacing in cases of pacemaker-dependence. For each patient, three maps will be created with the EnSite TurboMap Mapping Tool (Abbott, MN): 1) The voltage map; 2) The local activation time (LAT) map (activation map) and 3) The repolarization map. Bipolar electrograms were filtered at 30-300 Hz, noise filters on and unipolar electrograms were filtered at 0.5-100 Hz, noise filters on, as previously described. All EGMs will be analyzed offline using digital calipers on EnSite Cardiac Mapping System, (Abbott Labs, Abbott Park, IL, USA) by two independent physicians. Discrepancies will be adjudicated by a third independent physician. The maps will be manually edited to remove outliers LAT or RT points and if there was any doubt about the end of the repolarization the point will be removed from analysis. Scar will be defined as bipolar voltage <0.5mV and border zone will be defined as bipolar voltage 0.5 mV-1.5mV.

The LAT map will be performed using the LATlatest method, as recently described. Briefly, LATlatest will be annotated on: 1) the offset of the local high-frequency bipolar EGM potential, or 2) for EGMs with double potentials or LPs, the annotation will be at the offset of the second potential or LP, respectively. Each LAT map will be divided into 8 isochrones of activation. DZs will be defined as an area with >3 isochrones within 10 mm, as previously described.

The repolarization map will be performed using unipolar electrograms with the Wyatt method. Repolarization time (RT) will be defined as the time from the reference (onset of the surface QRS in ECG lead II) to the steepest positive dV/dT (maximum +dV/dT) of the unipolar T wave, as previously described. A steep repolarization gradient, an expression of heterogeneity, will be defined as "repolarization cliff" and determined if the time difference (∆) in RT between two neighboring regions within 1 cm distance is higher than a prespecified cutoff. In particular, a repolarization cliff will be defined as ∆RT>100 ms, based on previous studies.

FOLLOW-UP Patients will be followed up in the outpatient clinic every 6 months and by ICD remote monitoring. ICD implanted patients will also undergo serial device interrogations every 6 months. Primary endpoint will be VT recurrence after ablation, defined as: appropriate ICD therapy or monomorphic VT recurrence.

STATISTICAL ANALYSIS All variables will be tested for normality with Shapiro-Wilk test. Normally distributed variables will be described as mean ± standard deviation and the groups compared through paired or unpaired t-test as appropriate, while the non-normally distributed variables will be described as median (Inter Quartile Range) and compared by Mann-Whitney test as appropriate. The categorical variables will be described as frequencies (percentages) and compared by Chi-squared test or Fisher's exact test as appropriate. Cohen's kappa test will be used to assess interobserver agreement in EAM analysis.

A p-value less than 0.05 will be considered statistically significant. The analysis will be performed using R software version 3.6.2 (R Foundation for Statistical Computing, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

1. Ventricular tachycardia ablation procedure;
2. High density endocardial or epicardial substrate EAM performed with the multipolar mapping catheter Advisor™ HD-Grid Mapping Catheter, (Abbott Labs, Abbott Park, IL, USA) in association with the EnsiteXTM Cardiac Mapping System, (Abbott Labs, Abbott Park, IL, USA); 3) Use of TactiFlexTM ablation catheter (Abbott Labs, Abbott Park, IL, USA).

Exclusion Criteria:

1) use of a different mapping system

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients undergoing VT ablation at Universitair Ziekenhuis Brussel (UZB), Brussels, Belgium will be prospectively enrolled if inclusion criteria will be fulfilled. Inclusion criteria will be: 1) VT ablation procedure; 2) High density endocardial or epicardial substrate EAM performed with the multipolar mapping catheter Advisor™ HD-Grid Mapping Catheter, (Abbott Labs, Abbott Park, IL, USA) in association with the EnsiteXTM Cardiac Mapping System, (Abbott Labs, Abbott Park, IL, USA); 3) Use of TactiFlexTM ablation catheter (Abbott Labs, Abbott Park, IL, USA).
  Exclusion criteria will be: 1) use of a different EAM mapping system. Clinical VT will be defined as a VT that occurs spontaneously based on analysis of 12-lead ECG QRS morphology, following current guidelines. Sustained VT will be defined as lasting more than 30 s
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy outcome | 1 Year
  Primary endpoint will be VT recurrence after ablation, defined as: appropriate ICD therapy or monomorphic VT recurrence.

IPD SHARING:
Plan to Share IPD: No